CLINICAL TRIAL: NCT01822678
Title: Efficacy and Safety of Eslicarbazepine Acetate (BIA 2 093) in Acute Manic Episodes Associated With Bipolar I Disorder in a Double Blind, Randomised, Dose Titration, Placebo Controlled, Multicentre Clinical Trial
Brief Title: Efficacy and Safety of Eslicarbazepine Acetate (BIA 2-093) in Acute Manic Episodes Associated With Bipolar I Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIA-2093-203
Record Dates: First submitted 2013-03-28; First posted 2013-04-02 (Estimated); Results first posted 2013-08-02 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-02

CONDITIONS: Bipolar I Disorder
MeSH Terms: interventions — eslicarbazepine acetate; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Group 1: Eslicarbazepine Acetate, starting with 800 mg per day and up-titrated in 800 mg steps until 2400 mg (maximum dose) according to clinical response.
  Interventions: Drug: Eslicarbazepine Acetate
- Group 2 (Experimental): Group 2: Eslicarbazepine Acetate, starting with 600 mg per day and up-titrated in 600 mg steps until 1800 mg (maximum dose) according to clinical response.
  Interventions: Drug: Eslicarbazepine Acetate
- Group 3 (Placebo Comparator): Group 3: Placebo (change in daily number of tablets administered, according to clinical response).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eslicarbazepine Acetate — Eslicarbazepine Acetate, starting with 800 mg per day and up-titrated in 800 mg steps until 2400 mg (maximum dose) according to clinical response.
  Other Names: Eslicarbazepine Acetate tablets
  Arms: Group 1
Drug: Eslicarbazepine Acetate — Eslicarbazepine Acetate, starting with 600 mg per day and up-titrated in 600 mg steps until 1800 mg (maximum dose) according to clinical response.
  Other Names: Eslicarbazepine Acetate tablets
  Arms: Group 2
Drug: Placebo — Placebo
  Other Names: sugar pill
  Arms: Group 3

SUMMARY:
Multicentre, double-blind, randomised, parallel-group, placebo-controlled dose-titration study; depending on clinical efficacy, up-titration of dosage 3 and 6 days after start of treatment; maintenance of individual maximum dose for the rest of the total 3-week treatment period; subsequently, down-titration (according to the dose steps and the time intervals of up-titration) and administration of an established anti-manic therapy during the tapering-off period (in patients who discontinued treatment) or entry into a recurrence prevention study (Protocol PRA+SCO/BIA-2093-205; reported under separate cover) as an option for patients who responded to the study treatment

DETAILED DESCRIPTION:
Objectives:

The primary objective was to evaluate the dose-dependent efficacy of 2 dose-titration regimens of Eslicarbazepine Acetate (ESL) compared with placebo as therapy in patients with acute mania.

The secondary objective was to evaluate the safety and tolerability of 2 dose-titration regimens of Eslicarbazepine Acetate in comparison to placebo.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 years;
* a documented diagnosis of bipolar I disorder according to the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) criteria (i.e., 296.0, 296.4 or 296.6) [8];
* currently displaying an acute manic (including mixed) episode according to the DSM-IV criteria;
* a Young Mania Rating Scale (YMRS) total score of ≥20;
* symptoms of the current manic episode starting within 2 weeks prior to randomisation (V2, Day 1);
* able to undergo a standard evaluation, including clinical interview, ratings and laboratory studies;
* signed informed consent form;
* post-menopausal or otherwise incapable of becoming pregnant by reason of surgery or tubal ligation; women of childbearing potential had to present a serum pregnancy test consistent with a non-gravid state and had to use double-barrier contraception until the post-study visit (PSV).

Exclusion Criteria:

* a history of schizophrenia or schizoaffective disorder, psychotic features or rapid cycling;
* currently treated with carbamazepine or oxcarbazepine;
* a history of unresponsiveness, intolerance or hypersensitivity to related compounds (carbamazepine, oxcarbazepine or licarbazepine);
* use of any depot-neuroleptics for the current manic episode;
* abuse of stimulating drugs or use of any systemic sympathicomimetic drug within the previous 2 weeks;
* electroconvulsive therapy within the previous 3 months;
* a history of dependence or chronic abuse from alcohol, drugs or medications within the last year;
* judged clinically to be at risk of harm to self or others;
* second or third-degree atrioventricular blockade not corrected with a pacemaker;
* relevant electrocardiogram (ECG) or laboratory abnormalities;
* calculated creatinine clearance <30 mL/min [men: (140-age) x weight / serum creatinine x 72; women: (0.85) (140-age) x weight / serum creatinine x 72. Age in years, weight in kg, and serum creatinine in mg/dL];
* pregnant or nursing;
* participating in another drug clinical trial within the last 2 months before the randomisation visit;
* not ensured capability to perform the trial or to comply with the study protocol (e.g., mental retardation or severe inability to communicate);
* any other uncontrolled clinically relevant disorder;
* previous treatment with Eslicarbazepine Acetate;
* a history or presence of bone marrow impairment or depression (introduced by protocol amendment No. 1);
* a history or presence of acute intermittent porphyria (introduced by protocol amendment No. 1).

Patients receiving treatment for bipolar disorder or other central nervous system disorders at randomisation were excluded from randomisation. If the patients had previously used such medications the following restrictions had to be taken into account:

* Patients treated with bipolar disorder preventive medication (for carbamazepine or oxcarbazepine see exclusion criteria), antidepressants, antipsychotic, anxiolytic, antiparkinsonian, and/or other potentially centrally acting drugs had to be washed-out for at least 2 days prior to randomisation (V2, Day 1).
* Patients treated with lithium or valproate could only be randomised with plasma levels < 0.5 mmol/L and < 50 mg/L, respectively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2005-12; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrício Soares-da-Silva, MD, PhD, Study Director — BIAL - Portela & Ca. SA

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study centres: 23 centres: 2 centres in Austria, 6 centres in Czech Republic, 6 centres in Slovakia, 1 centre in Portugal, and 8 centres in Romania.
  First patient enrolled: 02 December 2005 Last patient completed: 23 November 2006
Pre-assignment Details: Patients who met the selection criteria at the randomisation visit (visit 2, Day 1) were randomised to 1 of the 3 treatment groups
Groups:
- ESL 800 mg: Group 1: Eslicarbazepine Acetate, starting with 800 mg per day and up-titrated in 800 mg steps until 2400 mg (maximum dose) according to clinical response.
  Eslicarbazepine Acetate : Eslicarbazepine Acetate, starting with 800 mg per day and up-titrated in 800 mg steps until 2400 mg (maximum dose) according to clinical response.
- ESL 600 mg: Group 2: Eslicarbazepine Acetate, starting with 600 mg per day and up-titrated in 600 mg steps until 1800 mg (maximum dose) according to clinical response.
  Eslicarbazepine Acetate : Eslicarbazepine Acetate, starting with 600 mg per day and up-titrated in 600 mg steps until 1800 mg (maximum dose) according to clinical response.
- Placebo: Group 3: Placebo (change in daily number of tablets administered, according to clinical response).
  Placebo : Placebo, sugar pill
Period: Overall Study
Arm/Group | ESL 800 mg | ESL 600 mg | Placebo
Started | 57 | 64 | 40
Treated | 57 | 64 | 40
Safety Population | 57 | 64 | 40
Intention-to-Treat Population (ITT) | 57 | 63 (1 patient was excluded from the ITT population because he did not have post baseline efficacy data) | 40
Per Protocol Population | 45 | 52 | 34
Completed | 45 | 49 | 29
Not Completed | 12 | 15 | 11
Not completed — Withdrawal by Subject | 5 | 4 | 4
Not completed — Adverse Event | 4 | 3 | 1
Not completed — Lack of Efficacy | 3 | 6 | 5
Not completed — Lost to Follow-up | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Demographic characteristics of patients (Safety population)
Groups:
- BIA 2-093 - 2400 mg (Maximum Dose): Group 1: Eslicarbazepine Acetate, starting with 800 mg per day and up-titrated in 800 mg steps until 2400 mg (maximum dose) according to clinical response.
  Eslicarbazepine Acetate : Eslicarbazepine Acetate, starting with 800 mg per day and up-titrated in 800 mg steps until 2400 mg (maximum dose) according to clinical response.
- BIA 2-093 - 1800 mg (Maximum Dose): Group 2: Eslicarbazepine Acetate, starting with 600 mg per day and up-titrated in 600 mg steps until 1800 mg (maximum dose) according to clinical response.
  Eslicarbazepine Acetate : Eslicarbazepine Acetate, starting with 600 mg per day and up-titrated in 600 mg steps until 1800 mg (maximum dose) according to clinical response.
- Total: Total of all reporting groups
Arm/Group | BIA 2-093 - 2400 mg (Maximum Dose) | BIA 2-093 - 1800 mg (Maximum Dose) | Placebo | Total
Number analyzed (Participants) | 57 | 64 | 40 | 161
Age, Customized [Number; unit: participants]
  18 - 20 Years | 2 (19.3) | 0 (14.3) | 0 (22.5) | 2 (12.98)
  20 - 30 Years | 9 (70.2) | 10 (76.2) | 9 (67.85) | 28 (12.79)
  30 - 40 Years | 15 (10.5) | 17 (9.5) | 8 (10.0) | 40 (13.19)
  40 - 50 Years | 15 | 16 | 11 | 42
  50 - 60 Years | 10 | 15 | 8 | 33
  60 - 70 Years | 6 | 5 | 3 | 14
  70 - 80 Years | 0 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 36 | 18 | 81
  Male | 30 | 28 | 22 | 80

OUTCOME MEASURES:

1. Primary Outcome: Change in the Young Mania Rating Scale (YMRS) Total Score at the End of the 3-week Treatment Period, in Relation to the Baseline.
Description: The YMRS is used to assess disease severity in patients who have been previously diagnosed with mania and it has proven psychometric properties through 11 item multiple-choice diagnostic questionnaire and the total score is determined from the summation of each 11 individual scores (and can range from 0 - 60) based on the patient's subjective feedback of his clinical condition over the previous 48 hours. A higher score indicates a worse rating for symptoms related to mania. At every visit throughout the study, investigators administered the YMRS. The results of the primary analysis of efficacy were calculated using Analysis of covariance (ANCOVA) with Last Observation Carried Forward (LOCF). Primary variable is presented through ANCOVA results for absolute change in YMRS total score from baseline (V2) to end of treatment (V7). A responder has at least 50% improvement (reduction) in the YMRS total score or has a total score of less than 12 points at the end of treatment period.
Time Frame: baseline and 3-week
Population: The ITT efficacy population consisted of all randomised patients who received at least one dose of investigational product and at least 1 post-baseline YMRS assessment. If a patient discontinues before the end of the 3-week treatment period then the last observation will be carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BIA 2-093 - 2400 mg (Maximum Dose) | BIA 2-093 - 1800 mg (Maximum Dose) | Placebo
Number analyzed (Participants) | 57 | 63 | 40
units on a scale | -14.2 (1.17) | -12.5 (1.12) | -10.3 (1.40)

ADVERSE EVENTS:
Time Frame: Up to 4 weeks
Description: Participants were followed for the duration of drug administration, an average of 4 weeks (titration and maintenance) plus up to 6 days (tapering-off, i.e. downtitration conducted on an individual basis corresponding to up-titration)
Arm/Group | BIA 2-093 - 2400 mg (Maximum Dose) | BIA 2-093 - 1800 mg (Maximum Dose) | Placebo
Serious Adverse Events (participants affected / at risk) | 2/57 | 2/64 | 1/40
Other Adverse Events (participants affected / at risk) | 20/57 | 25/64 | 10/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIA 2-093 - 2400 mg (Maximum Dose) (N=57) | BIA 2-093 - 1800 mg (Maximum Dose) (N=64) | Placebo (N=40)
Mania (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIA 2-093 - 2400 mg (Maximum Dose) (N=57) | BIA 2-093 - 1800 mg (Maximum Dose) (N=64) | Placebo (N=40)
Headache (Nervous system disorders) | 5 (5) | 7 (7) | 0 (0)
Dizziness (Nervous system disorders) | 5 (5) | 6 (6) | 4 (4)
Nausea (General disorders) | 4 (4) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (4) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0)
Agitation (Psychiatric disorders) | 2 (2) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other